CLINICAL TRIAL: NCT03131271
Title: Effect of Ice Bag Application to Femoral Region on Pain in Patients Undergoing Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut Bayındır, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TYL-2013-4765
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Percutaneous coronary intervention; Femoral arterial catheter; Pain; Cold application; Nursing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the experimental group, the researcher provided a cold application for 20 minutes by placing an ice bag to the site of the femoral catheter. Immediately after its removal, the responsible nurse removed the catheter. A neutral instruction set was used on each patient prior to application of the ice pack. Patients in the experimental group were told that they may or may not experience pain during the catheter removal. The patients were also told that the aim of the study was to measure the effect of ice bag application upon pain during catheter removal, and that ice pack application may or may not be effective in terms of their own pain.
  Interventions: Other: cold application
- Control Group (No Intervention): The control group received the standard clinic procedure in that the catheter was removed by the assigned nurse without any cold application to the femoral region. Each control patient was informed that some patients may experience pain during catheter removal, and that they may or may not experience pain. Patients were also told that their pain levels would be measured during catheter removal.

INTERVENTIONS:
Other: cold application — In the experimental group, the researcher provided a cold application for 20 minutes by placing an ice bag to the site of the femoral catheter.
  Arms: Experimental Group

SUMMARY:
Background: Removal of femoral arterial catheter causes pain, and current interventions used for reducing this pain are not sufficiently effective.

Aims: The aim of this study is to determine the pain reduction effectiveness of ice bag applications to the femoral region in patients undergoing percutaneous coronary intervention.

Design: A randomized controlled trial with repeated measures and two-group design.

Setting: This study was conducted at the Yilmaz-Mehmet Oztaskın Heart and Vascular Hospital located in Kayseri, Turkey.

Participants: The study was completed with a total of 104 patients who met the inclusion criteria: 52 each in the experimental group and the control group.

Methods: The data were collected by the researcher using Patient Identification Form, Numerical Rating Scale (NRS), and Vital Signs Monitoring Form. An ice bag was applied to patients in the experimental group for 20 minutes before removal of the catheter. The nurse performing the application was also responsible for the catheter removal, immediately after the ice bag was removed. Standard procedures of the clinic were applied to the control group. According to the relevant standard procedures, the catheter was removed by the nurse without making any other application to femoral region, and pressure was applied on catheter site. The pain experienced by the patients was evaluated before, and during removal and again while the nurse applied pressure on the catheter site after removal. The NRS scores were identified as NRS1, NRS2 and NRS3 for the three assessment, respectively.

DETAILED DESCRIPTION:
Although several arterial access routes may be employed during percutaneous coronary intervention (PCI), the femoral arterial site has been the most commonly used (1). However, during femoral artery interventions, many patients experience pain and discomfort during the removal of catheters previously inserted into the femoral region (2,3). Previous literature also provides evidence that both vasovagal responses and local vascular complications may develop when the pain induced by catheter removal is not effectively controlled (3-5); therefore, it is important to reduce the pain experienced by patients undergoing this procedure (6).

Pain caused by the removal of a femoral catheter may be controlled by using pharmacological methods such as treatment with morphine sulfate or lidocaine infiltration (2,3). However, it is also been observed that such approaches may cause complications such as increased bleeding, laceration of catheters, infection and temporary nerve injury (7-9). Pain may be also be controlled using non-pharmacological methods, which are patient-specific and aim to establish empathic communication with healthcare staff (10-13). Non-pharmacological methods used for pain control provided positive effects such as reduced anxiety and psychological support; notably, patients have expressed satisfaction with such non-pharmacological methods (14).

Cold application is a non-pharmacological method of pain control (6). Being one of the oldest and easiest forms of treatment, cold-application increases the threshold of pain and reduces the conduction velocity of nerve fibres transmitting pain stimuli from the peripheral to the central nervous system (15). Demir et al. (10) investigated the effect of cold application upon pain caused by the removal of a chest tube and revealed that cold application reduced pain intensity and delayed patient requests for a second analgesic. In a further study by Ertug et al. (11), cold application was highly effective in reducing the pain caused by chest tube removal. Cold application also confers other advantages, such as ease of application, the lack of serious side effects and low cost (16).

Aim and Hypothesis of the Study This study aimed to determine the effect of cold application to the femoral region upon pain levels of patients receiving PCI. Our hypothesis was that cold application would reduce (1) the pain score associated with removal of a femoral catheter after PCI, (2) the behavioural responses of discomfort associated with removal of a femoral catheter after PCI and (3) the incidence of adverse reactions associated with removal of a femoral catheter after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: able to speak and understand Turkish, over 18 years of age, about to undergo a femoral intervention to insert a single catheter in their femoral region, unimpaired time and place orientation with no psychiatric disorders or no visual or hearing problem, no cold allergy, normal vital signs and avoidance of analgesic treatment prior to catheter removal.

Exclusion Criteria:

* The exclusion criteria were; refusal to participate, groin lesion at the time of sheath removal, unstable vital signs, the use of radial acces

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | 9 months
  self reported pain intensity immediately prior to catheter removal, during catheter removal, and while the nurse applied pressure on catheter site within the first minute after removal

IPD SHARING:
Plan to Share IPD: No